CLINICAL TRIAL: NCT01038076
Title: Implementing Computerized Clinical Assessment of HIV Patient Adherence
Brief Title: Medications for Chronic HIV: Education and Collaboration
Acronym: MedCHEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); VA Office of Research and Development (U.S. Federal Agency); VA Boston Healthcare System (U.S. Federal Agency); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); San Diego State University (Other); Tufts University (Other)
Responsible Party: Principal Investigator, Allen L. Gifford, Professor of Public Health and Medicine, Boston University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-26736; R01MH076911-02 (NIH)
Record Dates: First submitted 2009-12-19; First posted 2009-12-23 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections; Acquired Immunodeficiency Syndrome; Medication Adherence
Keywords: HIV; AIDS; adherence; antiretroviral; aCASI; HAART; Complementary Therapies; Adherence Care Manager
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MedCHEC Tablet Computer & Adherence Care (Experimental): Patients assigned to the intervention answer questions about their medication, medication-taking behavior and risks for non-adherence on the MedCHEC tablet touch-screen computer, which generates provider and patient reports. Patients may be referred to an Adherence Care Manager on the basis of the reports. In addition, patients will receive standard information about adherence.
  Interventions: Behavioral: MedCHEC Tablet Computer & Adherence Care
- Adherence Information Only (No Intervention): Patients assigned to the active comparator arm will receive standard information about adherence.

INTERVENTIONS:
Behavioral: MedCHEC Tablet Computer & Adherence Care — Patients answer questions about their medication, medication-taking behavior and risks for non-adherence on the MedCHEC tablet touch-screen computer, which generates patient and provider reports. Patients may be referred to an Adherence Care Manager on the basis of the reports.
  Other Names: HIV/Adhere; aCASI
  Arms: MedCHEC Tablet Computer & Adherence Care

SUMMARY:
This study will examine whether a computerized, self-administered assessment of patient medication adherence and health behaviors, plus support for adherence, improves the ability of clinicians to identify adherence problems and leads to better adherence.

DETAILED DESCRIPTION:
Antiretroviral medications are highly effective in controlling HIV, if patients adhere to the regimen. However, HIV medication adherence problems are very common, and evidence is clear that providers have great difficulty 'diagnosing' poor adherence accurately. If healthcare providers can identify patients with adherence problems, they can intervene to help patients overcome these problems and take their medications as prescribed, which can improve symptoms and quality and length of life. Both clinicians and HIV positive patients will be recruited to this study. Before each clinic visit, patients randomized to the intervention will be asked to answer questions about their medications, medication-taking behavior, and risk-factors for non-adherence on MedCHEC, a tablet touch-screen computer that generates provider and patient reports. We will give these reports to the provider and patient to assist with the clinical visit. Based on the MedCHEC-generated report, the patient may be referred to an Adherence Care Manager (ACM). The ACM will assist the patient in overcoming adherence barriers by telephone and in-clinic counseling. The study will evaluate the effects of this system on adherence and clinical care using both quantitative methods (randomized controlled trials of effects on adherence and providers' adherence estimates), and qualitative methods.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Confirmed HIV-positive
* On or newly starting antiretroviral medication for HIV
* Under treatment at one of the study sites
* Available by telephone

Exclusion Criteria:

* Clinically diagnosed by provider with significant cognitive impairment, or Mini-Mental Status Exam score less than or equal to 22
* Inability to read English
* Inability or refusal to use MedCHEC touch-screen computer
* Inability or refusal to use any form of electronic drug monitoring device (MEMS)
* Never available by telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 371 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Patient adherence to HIV medications, as measured by MEMS data, and by self-report questionnaires. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Allen L Gifford, M.D., Principal Investigator — Boston University School of Public Health and School of Medicine
Locations (3):
- United States (3):
  - VA Greater Los Angeles, Los Angeles, California
  - VA Boston, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided